CLINICAL TRIAL: NCT00236522
Title: A Multicenter, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of Levofloxacin 750 mg Once Daily for 5 Days Versus Levofloxacin 500 mg Once Daily for 10 Days in the Treatment of Acute Bacterial Sinusitis in Adults.
Brief Title: A Comparison of the Safety and Efficacy of Two Different Regimens of Levofloxacin in the Treatment of Acute Bacterial Sinusitis(Sinus Infection) in Adults.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002809
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Sinusitis
Keywords: sinus infection; acute bacterial sinusitis; sinusitis; bacterial sinus infection
MeSH Terms: conditions — Sinusitis | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of two antibiotic regimens in the treatment of acute bacterial sinusitis (sinus infection) in non-hospitalized adult patients. A 5-day course of 750 milligrams of levofloxacin given by mouth once daily will be compared to a 10-day course of 500 milligrams of levofloxacin given by mouth once daily.

DETAILED DESCRIPTION:
When treating sinus infections (sinusitis) caused by bacteria, the traditional duration of therapy is between 10 and 14 days. In this randomized, double-blind study, 5 days of 750 milligrams of levofloxacin given once daily will be compared to 10 days of 500 milligrams of levofloxacin in the treatment of non-hospitalized adult patients who have acute bacterial sinusitis. To prevent the study doctor, study staff and patients from knowing which study drug they are taking, all study drug will manufactured to look the same and patients on the 5-day regimen will be given placebo for the last 5 days of their participation in the study. Patients will have a sinus specimen collected at the first visit. Safety evaluations will be conducted. The objective of the study is to demonstrate that, in the treatment of acute bacterial sinus infections, a 5-day course of 750 milligrams of levofloxacin given once daily is at least as effective as a 10-day course of 500 milligrams of levofloxacin given once daily and is well tolerated.

Patients will take by mouth 750 milligrams levofloxacin capsules once daily for 5 days followed by placebo capsules once daily for 5 days, or 500 milligrams levofloxacin capsules once daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute bacterial sinusitis, defined by clinical signs and symptoms lasting for less than 28 days and the presence of visible nasal infection, and confirmed by computed tomography (CT) or standard sinus x-rays
* Two or fewer episodes of bacterial sinusitis within the preceding 12 months
* Willing to undergo maxillary sinus puncture or endoscopy

Exclusion Criteria:

* Chronic sinusitis
* Use of systemic antibiotics within the past 72 hours
* Presence or history of serious complications of sinusitis
* Surgery for treating sinusitis
* Required daily use of more than 20 milligrams of prednisone (oral steroid)
* Cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2002-10; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Clinical success (resolution of patient signs and symptoms) at the post-therapy visit.

SECONDARY OUTCOMES:
Microbiologic response at the post-therapy visit and safety evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Levofloxacin 750 mg Once Daily for 5 Days Versus Levofloxacin 500 mg Once Daily for 10 days in the Treatment of Acute Bacterial Sinusitis in Adults — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=490&filename=CR002809_CSR.pdf